CLINICAL TRIAL: NCT07295327
Title: Randomized and Comparative Clinical Study on the Lipid-lowering Efficacy and Tolerability of Two Food Supplements in Mild Hypercholesterolemia
Brief Title: Effect of Two Food Supplements on Lipid Profile in Patients With Mild Hypercholesterolemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYNACOL-METACOL-2025
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Food supplement
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cynacol (Experimental): Cynacol (developed by BioDue S.p.A.) is a dietary supplement containing, artichoke dry extract, naringin, Silybum marianum dry extract, flaxseed oil, vitamin E and sunflower oil.
  Interventions: Dietary Supplement: Cynacol
- Metacol (Active Comparator): Metacol (developed by BioDue S.p.A.) is a dietary supplement containing coenzyme Q10, monacolin k and flax seed oil.
  Interventions: Dietary Supplement: Metacol

INTERVENTIONS:
Dietary Supplement: Cynacol — Cynacol (developed by BioDue S.p.A.) containing, artichoke dry extract, naringin, Silybum marianum dry extract, flaxseed oil, vitamin E and sunflower oil, 2 capsules/day after dinner for 90 days
  Arms: Cynacol
Dietary Supplement: Metacol — Metacol (developed by BioDue S.p.A.) containing coenzyme Q10, monacolin k and flaxseed oil, 2 capsules/day after dinner for 90 days
  Arms: Metacol

SUMMARY:
The primary outcome is to evaluate the effect of Cynacol on the change in LDL-C levels compared to Metacol after 90 days of supplementation.

The secondary outcomes are to evaluate:

- the change of TC, non-HDL cholesterol (non-HDL-C), apolipoprotein B (apoB), Tg, HDL-C levels after 90 days of supplementation with Cynacol compared to Metacol. The safety outcome is collection of the adverse events not related, related or possibly related to the study products.

DETAILED DESCRIPTION:
In the screening visit subject's demographic data, medical history, co-morbidities and concomitant medication will be collected. Patients with documented hypercholesterolemia (LDL-C values between 115 and 190 mg/dl) will be evaluate. Blood sample analysis will be prescribed to be performed before the next visit for the evaluation of TC, HDL-C, Tg, apoB, fasting plasma glucose (FPG), creatinine, uric acid, alanine aminotransferase (ALT), aspartate aminotransferase (AST) and creatinine phosphokinase (CPK). At the baseline visit, a computerized medical record will be compiled where the following data will be recorded: vital signs [weight, height, BMI, systolic blood pressure (SBP) and diastolic blood pressure (DBP)] and the laboratory tests (TC, HDL-C, Tg, apoB, FPG, creatinine, uric acid, ALT, AST and CPK). The subjects will be randomized in one of the 2 groups to receive Cynacol or Metacol. A sufficient amount of study product for 90 days will be delivered. Standardized diet and physical activity advice will be prescribed. Blood sample analysis will be prescribed to be performed before the next visit for the evaluation of TC, HDL-C, Tg, apoB, FPG, creatinine, uric acid, ALT, AST and CPK. After 45 days of treatment, following blood samples collection, vital signs and laboratory tests will be recorded. Any adverse events eventually occurred will be collected. After 90 days of treatment, following blood samples collection, vital signs and laboratory tests will be recorded. Any adverse events eventually occurred will be collected. The primary outcome is to evaluate the effect of Cynacol on the change in LDL-C levels compared to Metacol after 90 days of supplementation.

The secondary outcomes are to evaluate:

- the change of TC, non-HDL cholesterol (non-HDL-C), apolipoprotein B (apoB), Tg, HDL-C levels after 90 days of supplementation with Cynacol compared to Metacol. The safety outcome is collection of the adverse events not related, related or possibly related to the study products.

ELIGIBILITY:
Inclusion Criteria:

* age between 35-70 years
* both genders
* LDL-C levels between 115 and 190 mg/dl
* subjects able to understand the informed consent and sign it before enrollment in the study

Exclusion Criteria:

* personal history of cardiovascular disease or equivalent risk factors
* Tg levels ≥ 400 mg/dl
* obesity [body mass index (BMI) ≥ 30 kg/m²]
* taking hypolipidemic drugs or supplements that affect lipid metabolism
* diabetes mellitus
* known thyroid, liver, kidney or muscle diseases
* any medical or surgical condition that makes patient compliance with the study protocol complex or inconsistent
* any known allergy or hypersensitivity to one or more components of the food supplements

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
LDL Cholesterol | 3 months
  The primary outcome is to evaluate the change in LDL-C levels after 90 days of supplementation with Cynacol compared to Metacol

SECONDARY OUTCOMES:
Lipid profile parameters different from LDL | three months
  to evaluate the variation of TC, non-HDL cholesterol (non-HDL-C), apolipoprotein B (apoB), Tg, HDL-C after 90 days of treatment with Cynacol compared to Metacol

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No